CLINICAL TRIAL: NCT06463951
Title: Study on the Synchrony and Reciprocity of Bodily Movements and Prosody Between Psychotherapist and Patient During Psychotherapy
Brief Title: Synchrony and Reciprocity of Body Movements and Prosody Between Psychotherapist and Patient
Acronym: RECiPROsody
Status: Recruiting | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Istituto di Gestalt HCC Italy - Centro Clinico e di Ricerca in Psicoterapia HCC Italy (Unknown)
Responsible Party: Principal Investigator, Giovanni Pioggia, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2024-006
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Relationship, Professional Patient
Keywords: psychotherapy; facial mimicry; fidgeting; relational synchrony

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects starting psychotherapy at the HCC Italy Clinical and Psychotherapy Research Center: The population that decides to undertake psychotherapy is diverse, including individuals of various ages, genders, socioeconomic backgrounds, and occupations. Motivations can vary widely, but often include management of mental disorders, relationship problems, stress, and personal growth. Despite existing barriers, a growing number of people are recognizing the importance of mental well-being and seeking professional support: increasing awareness and reduced stigma related to psychological symptoms are making psychotherapy an increasingly considered option for improving mental well-being and quality of life.
  Interventions: Other: Psychotherapy - Gestalt psychotherapy

INTERVENTIONS:
Other: Psychotherapy - Gestalt psychotherapy — Gestalt psychotherapy is an aesthetic-phenomenological approach that aims to improve self-awareness and integration by promoting emotional and relational well-being through what is happening in the present moment in the relationship with the therapist. The patient's current experiences are explored to better understand problems and behaviors and by promoting relational self-regulation

SUMMARY:
Modern psychotherapy focuses on co-regulation, where therapist and patient interactively manage emotions. This co-regulation is seen in nonverbal communication like facial expressions, gestures, and prosody (vocal pitchs). Studies show body movements and even skin conductance synchronize between patients and therapists during sessions.

The RECiPROsody project builds on this by using technology (cameras, sensors) to record and analyze these synchronies in psychotherapy sessions. This project aims to understand how this "attunement" between therapist and patient contributes to successful therapy.

Researchers will explore how patients and therapists interact using a mobile app that records video, audio, physiological signals (heart rate), and movements. Questionnaires will assess patient well-being and therapist experience.

By studying these micro-processes, RECiPROsody hopes to gain insights into how the therapeutic relationship develops, including the connections between physical reactions, nonverbal communication, and overall progress. This knowledge can improve psychotherapeutic techniques and highlight the importance of the nonverbal communication in therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between the ages of 20 and 60 years old who are referred to the HCC Italy Clinical and Psychotherapy Research Center

Exclusion Criteria:

* Patients under 20 years of age
* Presence of paranoid or psychotic symptoms
* Admissions to psychiatric Operative Units that have occurred within the last year since the start of psychotherapy at the HCC Italy Clinical and Psychotherapy Research Center

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients admitted to the HCC Italy Clinical and Psychotherapy Research Center and who meet the inclusion and exclusion criteria will be enrolled, after signing informed consent
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) | The questionnaire will be administered to patients pre-intervention, before the start of psychotherapy [T0] and 6 months after the start of psychotherapy [T1].
  CORE-OM is a 34-item self-administered questionnaire useful for assessing the outcome of psychological interventions. The CORE items relate to four domains: subjective well-being (4 items), symptoms/problems (12 items), functioning (12 items), and risk (6 items). Use of the CORE-OM provides useful insights by facilitating understanding of the patient's progress during the psychotherapeutic process. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time).
  The total score is calculated by adding the response values of all 34 items. The minimum score that can be achieved is 0 and the maximum 136, with higher scores indicating higher distress. Severity consists of six categories, characterizing respondents' psychological distress as either healthy (a score < 6), low-level (6-9), mild (10-14), moderate (15-19), moderate-severe (20-24) or severe (a score > 24).
Therapist Response Questionnaire (TRQ) | The questionnaire will be filled out by psychotherapists after the first 4 psychotherapy sessions and every 4 sessions.
  The TRQ is a clinician report of 79 items that measure a wide spectrum of thoughts, feelings, and behaviors expressed by therapists toward their patients, ranging from relatively specific feelings (e.g., "I feel bored in sessions with him/her") to complex constructs, such as projective identification (e.g., "More than with most patients, I feel like I've been pulled into things that I didn't realize until after the session was over").
  Items are derived by reviewing the clinical, theoretical, and empirical literature on countertransference and related variables, so that the instrument could be used comparably by therapists of any orientation. The clinicians assess each item on a 5-point Likert scale, ranging from 1 (not true) to 5 (very true). A total TRQ score was calculated by summing all 79 variables. The minimum score that can be achieved is 79 and the maximum 395. This TRQ total score was supposed to capture the general level of self-reported countertransference.
Aesthetic Relational Knowing of the Therapist (ARK-T) | The questionnaire will be filled out by psychotherapists after the first 4 psychotherapy sessions.
  The ARK-T scale is a 21-items measure of the therapist's aesthetic and field intuition during the psychotherapeutic process. It is composed by three main factors, "Bodily Awareness" (8 items), "Intuitive Resonance" (8 items), "Affective Empathy" (5 items). Each item is scored on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). The score could range from 21 to 105 and it could be correlate with the outcome of psychotherapy, or even with the measurement of relational factors such as the therapist's responsiveness, his or her self-compassion, and many other aspects developed within the various psychotherapeutic approaches. It will thus be possible to correlate this particular type of insight, to date little studied in the literature, with the effectiveness of psychotherapy, as well as with other aspects of the therapist's training and personality, e.g., personal psychotherapy, caring attitude toward self, ethics of responsivity toward the patient.
Clinical Outcomes in Routine Evaluation - Assessment (CORE-A) | The instrument will be filled out by the therapist after the first 4 sessions.
  The CORE-A allows for the collection of demographic data regarding patient, referral (date, first episode, relapse), patient's resources (family, financial condition), previous or ongoing treatment to ongoing drug treatments, on the severity of the disorder (4-point scale) and its duration (<6 months, 6-12 months, >12 months, recurrent), data on self- and heterolesive risk (4-point scale), on the outcome of the assessment (accepted psychotherapy, sent, etc.)
Clinical Outcomes in Routine Evaluation - End of therapy (CORE-E) | The instrument will be filled out by the therapist 6 months after the start of psychotherapy [T1].
  The CORE-E, also filled out by the therapist, collects data (comparable with the Assessment) on the type of psychotherapy performed, modality, frequency, mode of termination, reassessment of problems assessed at assessment and risk, assessment of contextual factors (motivation, therapeutic alliance, level of mentalization), benefits of therapy (e.g, insight capacity, expression of problems and moods, coping strategies, ability to make decisions, to ask for help, subjective well-being, symptoms, daily functioning, interpersonal relationships, possible drug therapy, and to agreements on possible follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Pioggia, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallese, V. (2009). Mirror neurons, embodied simulation, and the neural basis of social identification. Psychoanalytic Dialogues, 19(5), 519-536. https://doi.org/10.1080/10481880903231910
- [Background] Reinecke K.C.H., Dvoretska1 D., Joraschky P., Lausberg H. (2020). Fidgeting Behavior During Psychotherapy: Hand Movement Structure Contains Information About Depressive Symptoms. Journal of Contemporary Psychotherapy, 50:323-329 doi: 10.1007/s10879-020-09465-5
- [Background] Schore J., Schore A. (2008). Modern attachment theory: the central role of affect regulation in development and treatment. Clin. Soc. Work J. 36: 9-20. doi: 10.1007/s10615-007-0111-7
- [Background] Tschacher W, Meier D. Physiological synchrony in psychotherapy sessions. Psychother Res. 2020 Jun;30(5):558-573. doi: 10.1080/10503307.2019.1612114. Epub 2019 May 6. PMID 31060474
- [Background] Wampold, B.E., Imel, Z. E. (2015). The Great Psychotherapy Debate: The Evidence for What Makes Psychotherapy Work. Abingdom: Routledge.